CLINICAL TRIAL: NCT02309359
Title: A Phase IIb Multicenter, Randomized, Double-blind, Placebo-Controlled Dose-Range Finding Study of ALX-0061 Administered Subcutaneously in Combination With Methotrexate, in Subjects With Moderate to Severe Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: A Dose-Range Finding Study for ALX-0061 Combination Therapy in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0061-C201; 2014-003033-26 (EudraCT Number)
Record Dates: First submitted 2014-11-27; First posted 2014-12-05 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ALX-0061; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo q2w + MTX (Placebo Comparator): Placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  Interventions: Other: Placebo; Drug: Methotrexate
- ALX-0061 75 mg q4w + MTX (Experimental): ALX-0061 75 mg every 4 weeks + placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  Interventions: Biological: ALX-0061; Other: Placebo; Drug: Methotrexate
- ALX-0061 150 mg q4w + MTX (Experimental): ALX-0061 150 mg every 4 weeks + placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  Interventions: Biological: ALX-0061; Other: Placebo; Drug: Methotrexate
- ALX-0061 150 mg q2w + MTX (Experimental): ALX-0061 150 mg every 2 weeks + placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  Interventions: Biological: ALX-0061; Other: Placebo; Drug: Methotrexate
- ALX-0061 225 mg q2w + MTX (Experimental): ALX-0061 225 mg every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24.
  The last study drug administration was at the Week 22 visit.
  Interventions: Biological: ALX-0061; Drug: Methotrexate

INTERVENTIONS:
Biological: ALX-0061
  Arms: ALX-0061 150 mg q2w + MTX; ALX-0061 150 mg q4w + MTX; ALX-0061 225 mg q2w + MTX; ALX-0061 75 mg q4w + MTX
Other: Placebo
  Arms: ALX-0061 150 mg q2w + MTX; ALX-0061 150 mg q4w + MTX; ALX-0061 75 mg q4w + MTX; Placebo q2w + MTX
Drug: Methotrexate — Stable background dose of commercially available methotrexate (not provided by the Sponsor).

SUMMARY:
The purpose of this study is to assess the efficacy and safety of dose regimens of ALX-0061 administered subcutaneously (s.c.) in combination with methotrexate (MTX) to subjects with active rheumatoid arthritis (RA) despite MTX therapy, compared with placebo.

To assess the effects of ALX-0061 on quality of life, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of ALX-0061, and to define the optimal dose regimen for ALX-0061, based on safety and efficacy, for further clinical development.

DETAILED DESCRIPTION:
Subjects who completed the 24-week assessment period and achieved at least 20% improvement in swollen joint count (SJC) and/or tender joint count (TJC) at Week 24 of study ALX0061-C201 were invited to participate in an open-label extension (OLE) study ALX0061-C203 (NCT02518620), if the study was approved in their country and selection criteria were met.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for at least 6 months prior to screening, and American College of Rheumatology (ACR) functional class I-III
* Subjects treated with and tolerating MTX
* Active RA
* Others as defined in the protocol

Exclusion Criteria:

* Have been treated with disease-modifying antirheumatic drugs (DMARDs)/systemic immunosuppressives other than MTX.
* Have received approved or investigational biological or targeted synthetic DMARD therapies for RA less than 6 months prior to screening.
* Have a history of toxicity, non-tolerance, primary non-response or inadequate response to a biological therapy, or targeted synthetic DMARDs, for RA.
* Have received prior therapy blocking the interleukin-6 (IL-6) pathway, at any time.
* Others as defined in the protocol

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ablynx Clinical Department, Study Director — Ablynx, a Sanofi company
Locations (84):
- United States (22):
  - Investigator Site, Birmingham, Alabama
  - Investigator Site, Hemet, California
  - Investigator Site, La Palma, California
  - Investigator Site, Los Angeles, California
  - Investigator site, Los Angeles, California
  - Investigator Site, Ventura, California
  - Investigator Sites, Hialeah, Florida
  - Investigator Site, Homestead, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Miami Lakes, Florida
  - Investigator Site, Orlando, Florida
  - Investigator Site, Stockbridge, Georgia
  - Investigator Site, Overland Park, Kansas
  - Investigator Site, Monroe, Louisiana
  - Investigator Site, Worcester, Massachusetts
  - Investigator Site, Albuquerque, New Mexico
  - Investigator Site, Brooklyn, New York
  - Investigator Site, New York, New York
  - Investigator Sie, Charleston, South Carolina
  - Investigator Site, Myrtle Beach, South Carolina
  - Investigator Site, Memphis, Tennessee
  - Investigator Site, Mesquite, Texas
- Belgium (3):
  - Investigator Site, Brussels
  - Investigator Site, Ghent
  - Investigator Site, Liège
- Bulgaria (6):
  - Investigator Site, Pleven
  - Investigator Site, Plovdiv
  - Investigator Site 1, Rousse
  - Investigator Site 2, Rousse
  - Investigator Site, Sofia
  - Investigator Site, Varna
- Czechia (4):
  - Investigator Site, Brno
  - Investigator Site, Olomouc
  - Investigator Site, Prague
  - Investigator Site, Zlín
- Georgia (3):
  - Investigator Site, Tbilisi
  - Investigator Site 1, Tbilisi
  - Investigator Site 2, Tbilisi
- Germany (5):
  - Investigator Site, Bad Nauheim
  - Investigator Site, Berlin
  - Investigator Site, Cologne
  - Investigator Site, Frankfurt
  - Investigator Site, Hamburg
- Hungary (8):
  - Investigator Site, Baja
  - Investigator Site, Balatonfüred
  - Investigator Site, Békéscsaba
  - Investigator Site, Budapest
  - Investigator Site, Gyula
  - Investigator Site, Székesfehérvar
  - Investigator Site, Szikszó
  - Investigator Site, Veszprém
- Mexico (7):
  - Investigator Site, Culiacán
  - Investigator Site, León
  - Investigator Site 1, Mexico City
  - Investigator Site 2, Mexico City
  - Investigator Site, Mérida
  - Investigator Site, Monclova
  - Investigator Site, Monterrey
- Investigator Site, Chisinau, Moldova
- North Macedonia (2):
  - Investigator Site 1, Skopje
  - Investigator Site 2, Skopje
- Poland (10):
  - Investigator Site, Bydgoszcz
  - Investigator Site, Elblag
  - Investigator Site, Gdynia
  - Investigator Site, Grodzisk Mazowiecki
  - Investigator Site, Katowice
  - Investigator Site, Lublin
  - Investigator Site, Poznan
  - Investigator Site, Sochaczew
  - Investigator Site, Torun
  - Investigator Site, Warsaw
- Romania (5):
  - Investigator Site, Brăila
  - Investigator Site, Bucharest
  - Investigator Site, Oradea
  - Investigator Site, Târgu Mureş
  - Investigator Site, Timișoara
- Serbia (5):
  - Investigator Site 1, Belgrade
  - Investigator Site 2, Belgrade
  - Investigator Site 3, Belgrade
  - Investigator Site, Niška Banja
  - Investigator Site, Novi Sad
- Spain (3):
  - Investigator Site, Madrid
  - Investigator Site, Salamanca
  - Investigator Site, Santiago de Compostela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 345 subjects were recruited at 63 sites located in Europe (46 sites; 259 subjects), Latin America (7 sites; 59 subjects) and North America (10 sites; 27 subjects). Consent was obtained from the first subject on 30 Jan 2015; the last subject completed the final visit on 8 Aug 2016.
Pre-assignment Details: Of the 712 subjects screened, 367 were screen failures and 345 were randomly assigned to treatment (Intent-to-treat population). All subjects enrolled received study drug and were included in the safety population. All subjects who received at least one dose of ALX-0061 (i.e., 276 subjects) were included in the pharmacokinetic (PK) population.
Groups:
- ALX-0061 75 mg q4w + MTX: ALX-0061 75 mg every 4 weeks + placebo every 2 weeks + Methotrexate (MTX; at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  ALX-0061
  Placebo
  Methotrexate: Stable background dose of commercially available methotrexate (not provided by the Sponsor).
- ALX-0061 150 mg q4w + MTX: ALX-0061 150 mg every 4 weeks + placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  ALX-0061
  Placebo
  Methotrexate: Stable background dose of commercially available methotrexate (not provided by the Sponsor).
- ALX-0061 150 mg q2w + MTX: ALX-0061 150 mg every 2 weeks + placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  ALX-0061
  Placebo
  Methotrexate: Stable background dose of commercially available methotrexate (not provided by the Sponsor).
- ALX-0061 225 mg q2w + MTX: ALX-0061 225 mg every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24.
  The last study drug administration was at the Week 22 visit.
  ALX-0061
  Methotrexate: Stable background dose of commercially available methotrexate (not provided by the Sponsor).
- Placebo q2w + MTX: Placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  Placebo
  Methotrexate: Stable background dose of commercially available methotrexate (not provided by the Sponsor).
Period: Overall Study
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Started | 69 | 70 | 68 | 69 | 69
Completed | 57 | 62 | 57 | 57 | 60
Not Completed | 12 | 8 | 11 | 12 | 9
Not completed — Adverse Event | 4 | 5 | 5 | 4 | 4
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 4 | 0
Not completed — Lack of Efficacy | 3 | 1 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Other | 2 | 0 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- ALX-0061 75 mg q4w + MTX: ALX-0061 75 mg every 4 weeks + placebo every 2 weeks + MTX (at a stable dose and route) from baseline through Week 24. The last study drug administration was at the Week 22 visit.
  ALX-0061
  Placebo
  Methotrexate: Stable background dose of commercially available methotrexate (not provided by the Sponsor).
- Total: Total of all reporting groups
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX | Total
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 59 | 58 | 56 | 55 | 56 | 284
  >=65 years | 10 | 11 | 12 | 14 | 13 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.35) | 52 (13.16) | 51.9 (11.93) | 52.3 (13.36) | 52.8 (11.92) | 52.4 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 62 | 59 | 55 | 55 | 289
  Male | 11 | 8 | 9 | 14 | 14 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects Achieving American College of Rheumatology (ACR) 20 Response at Week 12
Description: ACR 20 response is defined as:
  * 20% improvement in tender joint count (TJC; 68 joints) relative to Week 0 AND
  * 20% improvement in swollen joint count (SJC; 66 joints) relative to Week 0 AND
  * 20% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - visual analogue scale [VAS])
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI)
    * C-reactive protein (CRP) level
  The primary endpoint was analyzed using non-responder imputation (NRI), i.e., subjects with missing ACR20 response at Week 12 were treated as non responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants | 52 | 57 | 53 | 50 | 43
Statistical Analysis 1: Comparison: ALX-0061 75 mg q4w + MTX vs ALX-0061 150 mg q4w + MTX vs ALX-0061 150 mg q2w + MTX vs ALX-0061 225 mg q2w + MTX vs Placebo q2w + MTX; The null hypothesis of this test was that there is no difference in the percentage of subjects achieving ACR20 response between the treatment groups and the alternative hypothesis was that the percentage of subjects achieving ACR20 response increases with increasing dose level; Test type: Other — Under the assumption of monotonicity, a Cochran-Armitage trend test was performed as the primary efficacy analysis. Data were analyzed according to the intent-to-treat (ITT) principle; thus, subjects were analyzed according to the treatment to which they were assigned. Subjects with missing ACR20 response at Week 12 were treated as non responders (non responder imputation approach); p = 0.172, Cochran-Armitage trend test

2. Secondary Outcome: Number and Percentage of Subjects With ACR20 Response at Week 24
Description: ACR 20 response is defined as:
  * 20% improvement in tender joint count (TJC; 68 joints) relative to Week 0 AND
  * 20% improvement in swollen joint count (SJC; 66 joints) relative to Week 0 AND
  * 20% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - visual analogue scale [VAS])
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI)
    * C-reactive protein (CRP) level
  This endpoint was analyzed using NRI, i.e., subjects with missing response at Week 24 were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants | 51 | 55 | 49 | 52 | 51

3. Secondary Outcome: Number and Percentage of Subjects With ACR50 Response at Weeks 12 and 24
Description: ACR50 response is defined as:
  * 50% improvement in TJC (68 joints) relative to Week 0 AND
  * 50% improvement in SJC (66 joints) relative to Week 0 AND
  * 50% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - VAS)
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by HAQ-DI
    * CRP level
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 20 | 31 | 28 | 31 | 19
  Week 24 | 33 | 39 | 37 | 42 | 27

4. Secondary Outcome: Number and Percentage of Subjects With ACR70 Response at Weeks 12 and 24
Description: ACR70 response is defined as:
  * 70% improvement in TJC (68 joints) relative to Week 0 AND
  * 70% improvement in SJC (66 joints) relative to Week 0 AND
  * 70% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - VAS)
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by HAQ-DI
    * CRP level
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 10 | 15 | 13 | 12 | 6
  Week 24 | 16 | 23 | 15 | 31 | 12

5. Secondary Outcome: Number and Percentage of Subjects With Low Disease Activity (LDA) Using Disease Activity Score 28 (DAS28) Using C-reactive Protein (CRP) at Weeks 12 and 24
Description: DAS28(CRP) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.36 × ln[CRP+1]) + (0.014 × VASPA) + 0.96
  Low disease activity = 2.6 ≤ DAS28 ≤ 3.2
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 16 | 37 | 32 | 40 | 16
  Week 24 | 26 | 40 | 41 | 48 | 20

6. Secondary Outcome: Number and Percentage of Subjects With LDA Using DAS28 Using Erythrocyte Sedimentation Rate (ESR) at Weeks 12 and 24
Description: DAS28(ESR) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.70 × ln[ESR]) +(0.014 × VASPA)
  Low disease activity = 2.6 ≤ DAS28 ≤ 3.2
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 13 | 36 | 29 | 33 | 11
  Week 24 | 24 | 38 | 33 | 46 | 13

7. Secondary Outcome: Number and Percentage of Subjects With LDA Using Simplified Disease Activity Index (SDAI) at Weeks 12 and 24
Description: SDAI = TJC28 + SJC28 + Patient's Global Assessment of Disease Activity (VASPA) + Physician's Global Assessment of Disease Activity (VASPHA) + CRP (mg/dL)
  Low disease activity: 3.3 < SDAI ≤ 11.0
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 49 | 34 | 29 | 25 | 17
  Week 24 | 29 | 34 | 35 | 46 | 22

8. Secondary Outcome: Number and Percentage of Subjects With LDA Using Clinical Disease Activity Index (CDAI) at Weeks 12 and 24
Description: CDAI = TJC28 + SJC28 + VASPA + VASPHA
  Low disease activity: 2.8 < CDAI ≤ 10
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 22 | 31 | 26 | 23 | 17
  Week 24 | 29 | 33 | 29 | 43 | 23

9. Secondary Outcome: Number and Percentage of Subjects With European League Against Rheumatism (EULAR) (CRP) Good Response at Weeks 12 and 24
Description: EULAR good response is defined as an improvement of >1.2 in DAS28 (CRP) relative to baseline.
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 15 | 36 | 30 | 39 | 15
  Week 24 | 26 | 39 | 39 | 47 | 19

10. Secondary Outcome: Number and Percentage of Subjects in Remission Using DAS28 (ESR) at Weeks 12 and 24
Description: DAS28(ESR) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.70 × ln[ESR]) +(0.014 × VASPA)
  Remission = DAS28(ESR) < 2.6
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 3 | 26 | 15 | 21 | 6
  Week 24 | 17 | 26 | 23 | 37 | 8

11. Secondary Outcome: Number and Percentage of Subjects in Remission Using SDAI at Weeks 12 and 24
Description: SDAI = TJC28 + SJC28 + VASPA + VASPHA + CRP (mg/dL)
  Remission: SDAI ≤ 3.3
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 2 | 8 | 6 | 5 | 3
  Week 24 | 7 | 13 | 10 | 14 | 6

12. Secondary Outcome: Number and Percentage of Subjects in Remission Using CDAI at Weeks 12 and 24
Description: CDAI = TJC28 + SJC28 + VASPA + VASPHA
  Remission: CDAI ≤ 2.8
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 3 | 7 | 4 | 5 | 3
  Week 24 | 10 | 13 | 8 | 13 | 7

13. Secondary Outcome: Number and Percentage of Subjects in Remission Using Boolean Defined Remission Criteria at Weeks 12 and 24
Description: Boolean remission: tender joint count (TJC)28 ≤ 1 and swollen joint count (SJC)28 ≤ 1 and VASPA (cm) ≤ 1 and CRP (mg/dL) ≤ 1
  This endpoint was analyzed using non-responder imputation (NRI), i.e., subjects with missing response at the concerned visit were treated as non responders.
Time Frame: 24 weeks
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Week 12 | 0 | 5 | 2 | 4 | 3
  Week 24 | 6 | 9 | 6 | 13 | 6

14. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Weeks 12 and 24
Description: The HAQ-DI is a 20-question instrument which assesses the degree of difficulty the subject had in accomplishing tasks in 8 functional areas over the previous week. The 8 areas are: dressing and grooming, hygiene, arising, reach, eating, grip, walking, common daily activities. Within each area, subjects report the amount of difficulty they have in performing the specific items. There are 4 response options ranging from: 0 = No Difficulty, 1 = With Some Difficulty, 2 = With Much Difficulty, 3 = Unable to Do. The 8 areas are each given a single score equal to the maximum value of their component activities (0, 1, 2, or 3). The sum of the area scores is then divided by the number of areas answered to obtain the final HAQ score (rounded to the nearest value evenly divisible by 0.125). The final HAQ-DI score ranges from 0 to 3. A high score means a high degree of disability (=worse outcome).
  Missing values were imputed with the last non-missing observation.
Time Frame: from baseline till Week 24
Population: Intent-to-treat population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
score on a scale
  Week 12 | -0.696 (0.0857) | -0.619 (0.0657) | -0.771 (0.0763) | -0.615 (0.0858) | -0.613 (0.0718)
  Week 24 | -0.82 (0.0913) | -0.665 (0.0682) | -0.876 (0.0802) | -0.772 (0.0926) | -0.662 (0.0798)

15. Secondary Outcome: Change From Baseline in Physical Component Score of Short Form Health Survey (SF-36) at Weeks 12 and 24
Description: The Short Form (36) Health Survey (SF-36) consists of 36 items that can be summarized into 8 domains: physical functioning, role limitations due to physical health problems (role-physical), bodily pain, general health, vitality, social functioning, role limitations due to emotional problems (role-emotional), and mental health. Two summary measures, the physical component summary and the mental component summary, can be derived based on these domain scores. Each score is directly transformed into a 0-100 score on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Time Frame: from baseline till Week 24
Population: Intent-to-treat population; "Number Analyzed" reflect the number of non-missing, non-imputed observations at that specific timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
score on a scale
  Week 12: number analyzed (Participants) | 61 | 66 | 58 | 60 | 59
  Week 12 | 7.372 (0.9136) | 7.100 (0.7477) | 6.534 (0.8878) | 7.778 (0.994) | 5.413 (0.7813)
  Week 24: number analyzed (Participants) | 58 | 62 | 58 | 58 | 59
  Week 24 | 10.412 (1.0642) | 8.725 (0.9194) | 8.835 (1.009) | 10.762 (1.1497) | 7.255 (0.9483)

16. Secondary Outcome: Change From Baseline in Mental Component Score of Short Form Health Survey (SF-36) at Weeks 12 and 24
Description: as for outcome 15
Time Frame: from baseline till Week 24
Population: as for outcome 15
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
score on a scale
  Week 12: number analyzed (Participants) | 61 | 66 | 58 | 60 | 60
  Week 12 | 9.096 (1.4966) | 7.249 (1.1237) | 9.749 (1.4177) | 5.686 (1.6485) | 5.569 (1.6467)
  Week 24: number analyzed (Participants) | 58 | 62 | 58 | 58 | 60
  Week 24 | 9.857 (1.5326) | 7.962 (1.3932) | 11.739 (1.4159) | 8.981 (1.6876) | 6.198 (1.696)

17. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Subscale at Weeks 12 and 24
Description: The FACIT Measurement System is a collection of health-related quality of life questionnaires that assess multidimensional health status in people with various chronic illnesses. The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: from baseline till Week 24
Population: as for outcome 15
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
score on a scale
  Week 12: number analyzed (Participants) | 61 | 65 | 58 | 61 | 60
  Week 12 | 11.014 (1.3593) | 8.63 (1.0465) | 10.884 (1.5424) | 9.389 (1.3706) | 6.381 (1.2026)
  Week 24: number analyzed (Participants) | 58 | 62 | 58 | 61 | 62
  Week 24 | 12.446 (1.5687) | 10.439 (1.2157) | 13.374 (1.5621) | 12.381 (1.5193) | 6.712 (1.4651)

18. Secondary Outcome: Pharmacokinetics: ALX-0061 Concentration in Serum at Weeks 12 and 24
Description: ALX-0061 concentrations were only measured in samples of subjects randomized to any of the ALX-0061 treatment arms. Samples were taken predose at the concerned visits.
Time Frame: at Week 12 and Week 24 visits
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69
micrograms/milliliter
  Week 12 | 0.163 (3.7) | 1.79 (3.08) | 19.9 (1.56) | 32.1 (1.43)
  Week 24 | 0.122 (2.56) | 1.64 (3.11) | 20.9 (1.5) | 35.2 (1.37)

19. Secondary Outcome: Pharmacodynamics: Concentrations of Soluble Interleukin-6 Receptor (sIL-6R) at Weeks 12 and 24
Description: Values below the limit of quantification are imputed with the lower limit of quantification (LLOQ).
Time Frame: from baseline till Week 24
Population: Safety Population; "Number Analyzed" reflect the number of subjects with data available at that specific timepoint.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
ng/mL
  Baseline | 26.9 (0.995) | 29.2 (1.04) | 27.7 (0.78) | 28.9 (1.05) | 28.9 (1.1)
  Week 12: number analyzed (Participants) | 62 | 66 | 57 | 61 | 60
  Week 12 | 166 (16.7) | 420 (21) | 519 (16.8) | 488 (16.8) | 52.9 (14.1)
  Week 24: number analyzed (Participants) | 58 | 61 | 58 | 59 | 60
  Week 24 | 150 (12.9) | 422 (17.8) | 484 (16.3) | 487 (14.3) | 35.4 (6.6)

20. Secondary Outcome: Number of Subjects With Development of a Treatment-emergent Antidrug Antibody Response
Time Frame: from baseline till follow-up (FU) (i.e., 12 weeks after last study drug dosing at Week 22 or after early treatment discontinuation)
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- ALX-0061 Total: All participants who received ALX-0061
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX | ALX-0061 Total
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69 | 276
Participants | 9 | 16 | 31 | 33 | 13 | 89

21. Secondary Outcome: Number and Percentage of Subjects With Treatment-emergent Adverse Events by Severity
Time Frame: From first study drug intake until the Week 24 or Early Termination visit. Only safety data through Week 24 is reported as 256 of the 293 subjects who completed the 24-week treatment period rolled-over to the C203 Study and did not perform the FU visit
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants
  Mild | 21 | 28 | 23 | 20 | 20
  Moderate | 15 | 12 | 19 | 20 | 14
  Severe | 6 | 4 | 2 | 4 | 2

22. Secondary Outcome: Number of Treatment-emergent Adverse Events by Severity
Time Frame: as for outcome 21
Population: Safety population
Measure: Number; unit: Adverse events
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Adverse events
  Mild | 66 | 78 | 66 | 56 | 49
  Moderate | 34 | 24 | 26 | 40 | 22
  Severe | 6 | 5 | 4 | 5 | 2

23. Secondary Outcome: Number and Percentage of Subjects With Treatment-related Treatment-emergent Adverse Events
Time Frame: as for outcome 21
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Participants | 26 | 25 | 26 | 25 | 18

24. Secondary Outcome: Number of Treatment-related Treatment-emergent Adverse Events
Time Frame: as for outcome 21
Population: Safety population
Measure: Number; unit: Adverse events
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
Number analyzed (Participants) | 69 | 70 | 68 | 69 | 69
Adverse events | 55 | 52 | 46 | 47 | 21

ADVERSE EVENTS:
Time Frame: From first study drug intake up to and including follow-up, i.e., maximum of 34 weeks (22 weeks of treatment + 12 weeks of follow-up).
Arm/Group | ALX-0061 75 mg q4w + MTX | ALX-0061 150 mg q4w + MTX | ALX-0061 150 mg q2w + MTX | ALX-0061 225 mg q2w + MTX | Placebo q2w + MTX
All-Cause Mortality (participants affected / at risk) | 1/69 | 0/70 | 0/68 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 5/69 | 5/70 | 0/68 | 2/69 | 4/69
Other Adverse Events (participants affected / at risk) | 29/69 | 34/70 | 27/68 | 38/69 | 17/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0061 75 mg q4w + MTX (N=69) | ALX-0061 150 mg q4w + MTX (N=70) | ALX-0061 150 mg q2w + MTX (N=68) | ALX-0061 225 mg q2w + MTX (N=69) | Placebo q2w + MTX (N=69)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0061 75 mg q4w + MTX (N=69) | ALX-0061 150 mg q4w + MTX (N=70) | ALX-0061 150 mg q2w + MTX (N=68) | ALX-0061 225 mg q2w + MTX (N=69) | Placebo q2w + MTX (N=69)
Hypertension (Vascular disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 2 (2) | 2 (2) | 6 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 5 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 4 (5) | 5 (7) | 7 (8) | 3 (3) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 4 (6) | 5 (6) | 4 (4)
Bronchitis (Infections and infestations) | 6 (7) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (5) | 2 (2) | 4 (4) | 6 (6)
Pharyngitis (Infections and infestations) | 2 (2) | 6 (6) | 3 (4) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 3 (3)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki, and will require prior review and written agreement of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT02309359/Prot_SAP_000.pdf